CLINICAL TRIAL: NCT05064826
Title: Measuring Improvement in the Quality of Emergency Department-initiated Treatment for Opioid Use Disorders Using Observation
Brief Title: ED Observation for Opioid Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01951; 19-A0-00-1002485 (Other Grant/Funding Number: nih)
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard visit (No Intervention): Participants will have standard Emergency Department visit as per standard operating procedures which should last approximately 3 -5 hours.
- Extended visit with Observation (Experimental): Participants will have extended Emergency Department visit by having an observation (which could be up to 23 hours) time in addition to the standard ED visit. In addition, information will be gathered about about the participants, use of opioids, healthcare visits, the quality of health, life, and treatment, and other topics. Urine or saliva or both may also be collected.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Emergency Department Observation Units (EDOU) would allow the highest risk patients - those presenting for nonfatal overdose - to receive their first dose of BUP before leaving the ED.
  Operationally defined to include placement in an observation unit and/or placement under observation status with care provided by Emergency Medicine and/or other services (e.g., Internal medicine, Psychiatry)
  Arms: Extended visit with Observation

SUMMARY:
This is a multicenter, randomized clinical comparative effectiveness trial (RCT) in which patients with untreated OUD presenting to a Northwell Health Emergency Department (ED), NYULH-Brooklyn, NYULH-Tisch, and Bellevue Hospital will be randomized (1:1) to be managed clinically through either a standard ED visit or an extended visit through ED observation (EDOU).

DETAILED DESCRIPTION:
In this hybrid implementation-effectiveness study, there is no direct research intervention. Rather, clinical care with well-documented effectiveness will be delivered at the discretion of clinical staff guided by clinical protocols for the management of OUD with MOUD (Medications for Opioid Use Disorder) introduced at each site prior to study enrollment. Enrolled patients will be randomized to ED vs. EDOU and to participate in assessments conducted at the index visit and at 30 days and 90 days. Patient level data will also be matched with Medicaid claims data for more robust analyses and to support the development of clinical quality measures.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or older
* Is able to speak English sufficiently to understand study procedures
* Has a history of non-medical opioid use
* Is a potential candidate for ED-based MOUD treatment initiation and referral at the site as confirmed by clinical staff
* s not receiving MOUD through ongoing formal addiction treatment or pain management at the time of index ED visit
* Is willing to receive either standard ED care or enhanced ED care in EDOU depending on random assignment
* Presents to the ED during study screening hours

Exclusion Criteria:

* Unwilling or unable to provide written/electronic informed consent/HIPAA Authorization for research procedures, including research visits at baseline and Day 30 and Day 90, and/or consent for the release of health records and data matching for a period of 2 years following enrollment and 1 year prior to enrollment.
* Currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or that could prevent participation in the study
* Presents from a medical-based extended care facility (e.g., skilled nursing facility)
* Previous participation in the current study
* Inadequate locator information (unable or unwilling to provide one unique mean of contact).
* Has acute, severe medical, psychiatric, or concurrent substance use problem or meets other criteria that would exclude the patient (clinically) from placement in EDOU according to EDOU placement clinical protocols.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who receive Emergency Department (ED)-initiated Buprenorphine (BUP) | Week 1 (~7-10 days)
  Receipt of ED-initiated BUP will be operationally defined to include administration of BUP and/or prescription for BUP as part of the ED/Emergency Department Observation (Units) (EDOU) visit. This measure will be abstracted from the health record primarily.
Proportion of participants who receive ED-initiated or ED-expedited BUP | Week 1 (~7-10 days)
  Receipt of ED-initiated/expedited BUP will be operationally defined to include the provision of a specific "warm" referral or transfer of care to a provider, clinic, or treatment setting with the capacity to administer and/or prescribe BUP within 24 hours of completion of the ED/EDOU visit. Eligible transition of care will be will described further in the Manual of Operations (MOP) and will include direct transport or handoff to an outpatient provider immediately from the ED, provision of an appointment within 24 hours (with a specific time and location), transfer to general inpatient or inpatient OUD/addiction treatment. Neither confirmation of a completed appointment (i.e., patient shows up and is seen) nor receipt of BUP at the dedicated follow-up appointment will be required as the patient and treating provider may elect to treat with alternative regimes (e.g., methadone, naltrexone). This measure will be abstracted from the health record primarily.
Proportion of participants who receive ED-initiated or ED-expedited Medications for Opioid Use Disorder (MOUD) | Week 1 (~7-10 days)
  Receipt of ED-initiated MOUD, inclusive of BUP, methadone, or naltrexone.
The proportion of participants who are successfully linked to formal addiction treatment within one week following the completion of their index ED/EDOU visit | Week 1 (~7-10 days)
  Successful linkage to formal addiction treatment will be defined as confirmed attendance at formal addiction treatment for OUD following completion of the ED/EDOU visit. Formal addiction treatment will be those treatments consistent with the American Society of Addiction Medicine's (ASAM) level of care (1-4) and will include a range of clinical settings, including office-based providers of BUP or naltrexone, Opioid Treatment Programs (OTPs), intensive outpatient, inpatient, or residential treatments. Means of confirmation will include direct contact with the facility and/or treating clinician or other objective means (e.g., medical record review).
The proportion of participants who are confirmed to be engaged in formal addiction treatment for OUD on the 30th day following the completion of their index ED/EDOU visit | Day 30
  Engagement in treatment for OUD will be defined as confirmed enrollment in formal addiction treatment for OUD on the 30th day following completion of the ED/EDOU visit. Attendance at two or more visits for formal addiction treatment within the 30-day period also constitutes engagement.

SECONDARY OUTCOMES:
Change in number of days of opioid and other drug use | Baseline, Day 30
  Measured by the Timeline Follow-Back (TLFB) procedure will be used to elicit the participant's self-reported use of illicit substances at baseline and throughout study participation.
Change in number of days of opioid and other drug use | Day 30, Day 90
  Measured by the Timeline Follow-Back (TLFB) procedure will be used to elicit the participant's self-reported use of illicit substances at baseline and throughout study participation.
Change in proportion of participants who tested positive for illicit opioids/substances | Baseline, Day 30
Change in proportion of participants who tested positive for illicit opioids/substances | Day 30, Day 90
Change in number of overdose events and risk behaviors | Baseline, Day 30
Change in number of overdose events and risk behaviors | Day 30, Day 90
Change in score on EuroQol-5 Dimensions (EQ-5D) Scale | Baseline, Day 30
  EuroQol-5 Dimensions (EQ-5D): The EuroQol is a structured interview that collects general health information applicable to a wide range of health conditions and treatment, providing a simple descriptive profile and a single index value for health status between 0 (dead) and 1 (full health).
Change in score on EuroQol-5 Dimensions (EQ-5D) Scale | Day 30, Day 90
  EuroQol-5 Dimensions (EQ-5D): The EuroQol is a structured interview that collects general health information applicable to a wide range of health conditions and treatment, providing a simple descriptive profile and a single index value for health status between 0 (dead) and 1 (full health).
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS-29) Scale | Baseline, Day 30
  Assessment of quality of life in seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) all assessed using the PROMIS-29 questionnaire. PROMIS-29 is scored on a T-score metric with a mean of 50 and a standard deviation of 10 in the U.S. general population, with a higher score representing more symptoms.
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS-29) Scale | Day 30, Day 90
  Assessment of quality of life in seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) all assessed using the PROMIS-29 questionnaire. PROMIS-29 is scored on a T-score metric with a mean of 50 and a standard deviation of 10 in the U.S. general population, with a higher score representing more symptoms.
Change in score on Patient Health Questionnaire (PHQ)-9 Scale | Baseline, Day 30
  The PHQ-9 is a 9-item instrument used for screening, diagnosing, monitoring and measuring the severity of depression. Each item is rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27. Scores are interpreted as follows: Minimal Depression: 0-4, Mild depression: 5-9, Moderate depression: 10-14, Moderately severe depression: 15-19, Severe depression: 20-27.
Change in score on Patient Health Questionnaire (PHQ)-9 Scale | Day 30, Day 90
  The PHQ-9 is a 9-item instrument used for screening, diagnosing, monitoring and measuring the severity of depression. Each item is rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27. Scores are interpreted as follows: Minimal Depression: 0-4, Mild depression: 5-9, Moderate depression: 10-14, Moderately severe depression: 15-19, Severe depression: 20-27.
Change in score on Treatment Effectiveness Assessment (TEA) Scale | Baseline, Day 30
  Treatment Effectiveness Assessment (TEA) scale is comprised of 4 questions about substance use, health, lifestyle, and community. Participants respond the questions on how they have improved in that area on a scale from 1 (not better at all) to 10 (very much better). Higher scores indicate overall improvement and effectiveness of treatment.
Change in score on Treatment Effectiveness Assessment (TEA) Scale | Day 30, Day 90
  Treatment Effectiveness Assessment (TEA) scale is comprised of 4 questions about substance use, health, lifestyle, and community. Participants respond the questions on how they have improved in that area on a scale from 1 (not better at all) to 10 (very much better). Higher scores indicate overall improvement and effectiveness of treatment.
Change in proportion of participants who reported treatment satisfaction | Baseline, Day 30
Change in proportion of participants who reported treatment satisfaction | Day 30, Day 90
Change in proportion of participants who reported changes in social determinants of health (e.g., homelessness, employment) | Baseline, Day 30
  Self reported by participants.
Change in proportion of participants who reported changes in social determinants of health (e.g., homelessness, employment) | Day 30, Day 90
  Self reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCormack, MD, Principal Investigator — NYU Langone Health
Locations (6):
- United States (6):
  - Rutgers University-University Hospital, Newark, New Jersey
  - NYULH-Brooklyn, Brooklyn, New York
  - Northwell Health - Long Island Jewish Medical Center, New Hyde Park, New York
  - Bellevue, New York, New York
  - NYULH-Tisch, New York, New York
  - Northwell Health - Staten Island University Hospital, Staten Island, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to ryan.mccormack@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT05064826/ICF_000.pdf